CLINICAL TRIAL: NCT01383824
Title: A Multi-centre, Prospective, Uncontrolled Post Market Clinical Follow-up Study (PMCFS) to Monitor the Survival and Performance of the Silent™ Hip in Subjects Requiring a Total Hip Replacement
Brief Title: A Multi-centre Study to Assess the Long-term Performance of the Silent Hip™ in Primary Total Hip Replacement Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Rationalization of the Silent Hip Prosthesis for business reasons only
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT09/02
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2014-08

CONDITIONS: Primary Arthritis; Secondary Arthritis
Keywords: Hip Replacement; Femoral Component

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silent™ Hip (Other): A short cementless, femoral component for use in total hip arthroplasty
  Interventions: Device: Silent™ Hip

INTERVENTIONS:
Device: Silent™ Hip — A short cementless, femoral component for use in total hip arthroplasty

SUMMARY:
The purpose of this study is to monitor the performance and of the Silent Hip™ in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria:

* Any subject deemed suitable to receive the Silent™ Hip in combination with the Pinnacle™ acetabular cup system, in accordance with all applicable Instructions For Use, should be considered for entry into this study.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition/co-morbidity or infection that would compromise their long-term participation and follow-up in this study.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship | 5 years post-surgery

SECONDARY OUTCOMES:
Oxford Hip Score | 6 weeks-6 mths
University of California Los Angeles (UCLA) Activity Score | 6 weeks-6 mths
EuroQol EQ-5D | 6 weeks-6 mths
Harris Hip Score | 6 weeks-6 mths
Radiographic analysis | pre-discharge
Oxford Hip Score | 2 years
Oxford Hip Score | 3 years
Oxford Hip Score | 4 Years
Oxford Hip Score | 5 years
Oxford Hip Score | 6 Years
Oxford Hip Score | 7 Years
Oxford Hip Score | 8 Years
Oxford Hip Score | 9 years
Oxford Hip Score | 10 Years
Oxford Hip Score | 11 Years
Oxford Hip Score | 12 Years
Oxford Hip Score | 13 Years
Oxford Hip Score | 14 Years
Oxford Hip Score | 15 Years
University of California Los Angeles (UCLA) Activity Score | 2 years
University of California Los Angeles (UCLA) Activity Score | 3 years
University of California Los Angeles (UCLA) Activity Score | 4 Years
University of California Los Angeles (UCLA) Activity Score | 5 Years
University of California Los Angeles (UCLA) Activity Score | 6 Years
University of California Los Angeles (UCLA) Activity Score | 7 Years
University of California Los Angeles (UCLA) Activity Score | 8 Years
University of California Los Angeles (UCLA) Activity Score | 9 years
University of California Los Angeles (UCLA) Activity Score | 10 Years
University of California Los Angeles (UCLA) Activity Score | 11 Years
University of California Los Angeles (UCLA) Activity Score | 12 Years
University of California Los Angeles (UCLA) Activity Score | 13 Years
University of California Los Angeles (UCLA) Activity Score | 14 Years
University of California Los Angeles (UCLA) Activity Score | 15 years
EuroQol EQ-5D | 2 Years
EuroQol EQ-5D | 3 Years
EuroQol EQ-5D | 4 Years
EuroQol EQ-5D | 5 Years
EuroQol EQ-5D | 6 years
EuroQol EQ-5D | 7 years
EuroQol EQ-5D | 8 Years
EuroQol EQ-5D | 9 Years
EuroQol EQ-5D | 10 Years
EuroQol EQ-5D | 11 Years
EuroQol EQ-5D | 12 Years
EuroQol EQ-5D | 13 Years
EuroQol EQ-5D | 14 Years
EuroQol EQ-5D | 15 Years
Harris Hip Score | 2 Years
Harris Hip Score | 5 Years
Harris Hip Score | 10 Years
Harris Hip Score | 15 Years
Radiographic analysis | 6 weeks - 6 mths
Radiographic analysis | 1 year
Radiographic analysis | 2 Years
Radiographic analysis | 5 Years
Radiographic analysis | 10 years
Radiographic analysis | 15 Years

CONTACTS AND LOCATIONS:
Locations (9):
- Sygehus Sønderjyllands, Sønderborg, Denmark
- Orthopädie Kupfalz, Speyer, Germany
- Orthopaedic Clinic University La Sapienza, Rome, Italy
- Spain (3):
  - Hospital Nisa Sevilla-Aljarafe, Seville
  - Hospital San Juan de Dios del Aljarafe, Seville
  - Hospital Santa Ángela De La Cruz, Seville
- United Kingdom (3):
  - Princess Alexandra Hospital, Harlow, Essex
  - The Rivers Hospital, Sawbridgeworth, Hertfordshire
  - Wrightington Hospital, Wrightington, Lancashire